CLINICAL TRIAL: NCT03714464
Title: Effect of Physical Form of Apples on Gastrointestinal Function and Satiety: a MRI Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A13102015 SoM SPMIC PhD
Record Dates: First submitted 2018-10-10; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2017-08

CONDITIONS: Gastrointestinal Symptoms
Keywords: Gastrointestinal physiology; Gastrointestinal response to sugars; gastrointestinal; MRI; stomach; small bowel; sorbitol; excess fructose; FODMAPs; colon

STUDY DESIGN:
Intervention Model Description: The intervention to be tested in this study is dietary intake of apples which are naturally high in fermentable carbohydrate. The investigators purchased the apples from a mainstream high street supermarket.
  The test meals consisted of whole apples (Meal A), apple puree (Meal B) and apple juice (Meal C)
Masking Description: Principal investigators and co-investigators were blinded when measuring gastric volumes, small bowel water content and colonic volumes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole Apple (Experimental): Participants will be given 350g of whole apple and 150 mls water to be consumed in 20 minutes.
  Serial MRI of gastrointestinal tract is done every 45 minutes from baseline until 315 minutes.
  Interventions: Other: Whole apples
- Apple Puree (Experimental): Participants will be given 384g of apple puree and 150 mls water to be consumed in 20 minutes.
  Serial MRI of gastrointestinal tract is done every 45 minutes from baseline until 315 minutes.
  Interventions: Other: Apple puree
- Apple Juice (Experimental): Participants will be given 338g of apple juice and 150 mls water to be consumed in 20 minutes.
  Serial MRI of gastrointestinal tract is done every 45 minutes from baseline until 315 minutes
  Interventions: Other: Apple Juice

INTERVENTIONS:
Other: Whole apples — 350 of whole apples containing 49g of available carbohydrate with 173ml water
  Arms: Whole Apple
Other: Apple puree — 384g of apple puree containing 44g of available carbohydrates with 224 ml water
  Arms: Apple Puree
Other: Apple Juice — 338g apple juice containing 46g of available carbohydrate with 260 ml water
  Arms: Apple Juice

SUMMARY:
Different physical form of apples had a significant effect on satiety and blood sugar levels which was shown in a 1977 study by Haber and his team (Haber et al.1977).It was suggested that , this effect was due to processing of the apples which modified the bioavailability of carbohydrate and fiber content.However this was not enough to explain the mechanistic effect of the apples. Within the last decade, the role of magenetic resonance imaging has been very promising in understanding gastrointestinal function and physiology. Recent MRI studies have measured changes in gastrointestinal volumes due to the effect of fermentable carbohydrates.

Apple contains fermentable carbohydrates or FODMAPs. They are known to be poorly absorbed in the small and exert an osmotic effect by increasing markedly small bowel water content in the intestinal lumen as demonstrated in imaging studies.(Murray et al 2014 and Placidi et al 2012). A reduction of FODMAPs in the diet of IBS sufferers has been found to alleviate functional gut symptoms demonstrated in several randomised controlled trials.

In order to fully understand the 1977 Haber study, the investigators would like to repeat the study using modern MRI methods in healthy volunteers and measure the volume changes in the stomach, small bowel and colon. In addition appetite and symptoms would also be investigated after ingesting each test meal.

DETAILED DESCRIPTION:
18 healthy volunteers will participate in this 3-way crossover study. They will attend one morning for each study, with the studies separated by approximately 1 week. We will measure breath hydrogen before the test meal, and after that approximately every hour for the next 5 h. We will also scan the subjects at baseline, immediately after the test meal and then approximately every hour for 5 hours postprandially. Subjects will be scanned on a research dedicated 1.5T MRI scanner. At baseline and every time the subjects come out of the MRI scanner we will ask them to rate their feelings of fullness, hunger and appetite as well their gastrointestinal symptoms on 100mm VAS scales. The subjects will be fed three types of Pink Lady apples test meals: whole apple, apple puree and apple juice. The apples will be sourced from supermarkets. The apple juice and apple puree will be prepared for this study by Campden BRI, a world famous food science research institute in Chipping Campden, UK. Each test meal will approximately provide 46g of available carbohydrate; 180kcal

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Able to give informed consent

Exclusion Criteria:

* Aversion to the test product
* Unable to eat whole fruit due to poor dentition or other reasons
* Pregnancy and lactation declared by candidate
* History declared by the candidate of pre-existing gastrointestinal disorder that may affect bowel function
* A positive diagnosis of irritable bowel syndrome based on the Rome III criteria questionnaire
* Reported history of previous resection of the oesophagus, stomach or intestine (excluding appendix)
* Intestinal stoma
* Any medical condition potentially compromising participation in the study e.g. diabetes mellitus, respiratory disease limiting ability to lie in the scanner
* Contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury
* Unable to limit alcohol intake to ≤ 35 units/ week and ≤ 8 units per day during trial and to avoid alcohol the day before each study day
* Unable to stop drugs known to alter GI motility including mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists for the duration of the study (Selective serotonin reuptake inhibitors and low dose tricyclic antidepressants will be recorded but will not be an exclusion criteria)
* Antibiotic or prescribed probiotic treatment in the past 8 weeks
* Inability to lie flat or exceed scanner limits of weight <120kg
* Poor understanding of English language
* Participation in night shift work the week prior to the study day. Night work is defined as working between midnight and 6.00 AM
* Participation in any medical trials for the past 3 months
* Alteration in habitual diet in the last 6 months
* Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol e.g. cognitive dysfunction, chaotic lifestyle related to substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Mean difference of small bowel water content (SBWC) in ml as measured by MRI from baseline to 315 minutes following ingestion of whole apple, apple puree and apple juice. | every 45 minutes from 0 minutes until 315 minutes
  Small bowel water content will be measured in mililitres (ml) using in house software for every 45 minutes. Difference in means will be compared using repeated measure ANOVA.

SECONDARY OUTCOMES:
Mean difference of gastric volume measured by MRI from baseline to 315 minutes minutes following ingestion of whole apple, apple puree and apple juice. | every 45 minutes from 0 minutes until 315 minutes
  Gastric volume in milliliters will be measured using MRI software every 45 minutes.Difference in means will be compared using repeated measure ANOVA.
Mean breath hydrogen measured from baseline to 315 minutes | every 45 minutes from 0 minutes until 315 minutes
  Breath hydrogen is measured in parts per million (ppm) using a breath hydrogen meter

OTHER OUTCOMES:
Difference in symptom severity | every 45 minutes from 0 minutes until 315 minutes for every intervention (whole apple, apple puree and apple juice)
  Symptom severity measured using a visual analogue scale with a rating from 0 to 100 measured in millimeters (mm)
Difference in appetite | every 45 minutes from 0 minutes until 315 minutes for every intervention (whole apple, apple puree and apple juice)
  Appetite ratings measured using a visual analogue scale with a rating from 0 to 100 to rate fullness, satiety, hunger and desire to eat.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, MD,FRCP, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shepherd SJ, Lomer MC, Gibson PR. Short-chain carbohydrates and functional gastrointestinal disorders. Am J Gastroenterol. 2013 May;108(5):707-17. doi: 10.1038/ajg.2013.96. Epub 2013 Apr 16. PMID 23588241
- [Background] Gibson PR, Shepherd SJ. Food choice as a key management strategy for functional gastrointestinal symptoms. Am J Gastroenterol. 2012 May;107(5):657-66; quiz 667. doi: 10.1038/ajg.2012.49. Epub 2012 Apr 10. PMID 22488077
- [Background] Barrett JS, Gearry RB, Muir JG, Irving PM, Rose R, Rosella O, Haines ML, Shepherd SJ, Gibson PR. Dietary poorly absorbed, short-chain carbohydrates increase delivery of water and fermentable substrates to the proximal colon. Aliment Pharmacol Ther. 2010 Apr;31(8):874-82. doi: 10.1111/j.1365-2036.2010.04237.x. Epub 2010 Jan 22. PMID 20102355
- [Background] Murray K, Wilkinson-Smith V, Hoad C, Costigan C, Cox E, Lam C, Marciani L, Gowland P, Spiller RC. Differential effects of FODMAPs (fermentable oligo-, di-, mono-saccharides and polyols) on small and large intestinal contents in healthy subjects shown by MRI. Am J Gastroenterol. 2014 Jan;109(1):110-9. doi: 10.1038/ajg.2013.386. Epub 2013 Nov 19. PMID 24247211
- [Background] Placidi E, Marciani L, Hoad CL, Napolitano A, Garsed KC, Pritchard SE, Cox EF, Costigan C, Spiller RC, Gowland PA. The effects of loperamide, or loperamide plus simethicone, on the distribution of gut water as assessed by MRI in a mannitol model of secretory diarrhoea. Aliment Pharmacol Ther. 2012 Jul;36(1):64-73. doi: 10.1111/j.1365-2036.2012.05127.x. Epub 2012 May 14. PMID 22582872
- [Background] Halmos EP, Power VA, Shepherd SJ, Gibson PR, Muir JG. A diet low in FODMAPs reduces symptoms of irritable bowel syndrome. Gastroenterology. 2014 Jan;146(1):67-75.e5. doi: 10.1053/j.gastro.2013.09.046. Epub 2013 Sep 25. PMID 24076059
- [Background] Ong DK, Mitchell SB, Barrett JS, Shepherd SJ, Irving PM, Biesiekierski JR, Smith S, Gibson PR, Muir JG. Manipulation of dietary short chain carbohydrates alters the pattern of gas production and genesis of symptoms in irritable bowel syndrome. J Gastroenterol Hepatol. 2010 Aug;25(8):1366-73. doi: 10.1111/j.1440-1746.2010.06370.x. PMID 20659225
- [Background] Staudacher HM, Lomer MC, Anderson JL, Barrett JS, Muir JG, Irving PM, Whelan K. Fermentable carbohydrate restriction reduces luminal bifidobacteria and gastrointestinal symptoms in patients with irritable bowel syndrome. J Nutr. 2012 Aug;142(8):1510-8. doi: 10.3945/jn.112.159285. Epub 2012 Jun 27. PMID 22739368
- [Background] Staudacher HM, Irving PM, Lomer MC, Whelan K. Mechanisms and efficacy of dietary FODMAP restriction in IBS. Nat Rev Gastroenterol Hepatol. 2014 Apr;11(4):256-66. doi: 10.1038/nrgastro.2013.259. Epub 2014 Jan 21. PMID 24445613
- [Background] Haber GB, Heaton KW, Murphy D, Burroughs LF. Depletion and disruption of dietary fibre. Effects on satiety, plasma-glucose, and serum-insulin. Lancet. 1977 Oct 1;2(8040):679-82. doi: 10.1016/s0140-6736(77)90494-9. PMID 71495
- [Background] Muir JG, Rose R, Rosella O, Liels K, Barrett JS, Shepherd SJ, Gibson PR. Measurement of short-chain carbohydrates in common Australian vegetables and fruits by high-performance liquid chromatography (HPLC). J Agric Food Chem. 2009 Jan 28;57(2):554-65. doi: 10.1021/jf802700e. PMID 19123815
- [Background] Marciani L, Wright J, Foley S, Hoad CL, Totman JJ, Bush D, Hartley C, Armstrong A, Manby P, Blackshaw E, Perkins AC, Gowland PA, Spiller RC. Effects of a 5-HT(3) antagonist, ondansetron, on fasting and postprandial small bowel water content assessed by magnetic resonance imaging. Aliment Pharmacol Ther. 2010 Sep;32(5):655-63. doi: 10.1111/j.1365-2036.2010.04395.x. PMID 20626735
- [Derived] Krishnasamy S, Lomer MCE, Marciani L, Hoad CL, Pritchard SE, Paul J, Gowland PA, Spiller RC. Processing Apples to Puree or Juice Speeds Gastric Emptying and Reduces Postprandial Intestinal Volumes and Satiety in Healthy Adults. J Nutr. 2020 Nov 19;150(11):2890-2899. doi: 10.1093/jn/nxaa191. PMID 32805050